CLINICAL TRIAL: NCT04899440
Title: An Experimental Clinical Study to Assess the Gingivitis and Plaque Reduction Efficacy of an Oral-Irrigator After Three Weeks of Use
Brief Title: Measuring Efficacy of an Oral-Irrigator After Three Weeks of Use
Status: Completed | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021043
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Subjects will proceed to an area separated from the examiner/examination area to receive supervised oral hygiene instructions and product usage instructions.
Oversight: Unapproved Device: Yes

ARMS (2):
- Test Regimen (Experimental): Oral Irrigator + Manual toothbrush + toothpaste Subjects will brush their teeth twice daily and will use the oral irrigator once in the evening daily
  Interventions: Device: Water Flosser
- Control Regimen (Sham Comparator): Manual toothbrush + toothpaste Subjects will brush their teeth twice daily
  Interventions: Other: Control

INTERVENTIONS:
Device: Water Flosser — A pressurized stream of water to reduce gingivitis and remove adherent plaque
  Arms: Test Regimen
Other: Control — No Oral Irrigator Control
  Arms: Control Regimen

SUMMARY:
The primary objective of this exploratory study is to evaluate the efficacy of an Oral Irrigator in the reduction of gingivitis compared to a negative control over a 3 week period by using the Modified Gingival Index and the Gingival Bleeding Index. The secondary objective is to evaluate the efficacy of an Oral Irrigator in the reduction of plaque compared to a negative control using the extended Turesky Modified Quigley-Hein Index (TQHPI) after 3 weeks of use.

DETAILED DESCRIPTION:
This is a single-center, examiner-blind, three (3) week, two (2) treatment, parallel group, randomized study design. Thirty (30) subjects who have shown evidence of gingivitis and plaque will be enrolled in this study. Subjects will be evaluated for gingivitis using the Modified Gingival Index (MGI) and the Gingival Bleeding Index (GBI) and evaluated for plaque using the Turesky Modified Quigley-Hein Plaque Index (TQHPI) at two (2) time points: Baseline and after three (3) weeks of product use. Qualified subjects will be stratified and randomly assigned to one of the two treatment groups, toothbrushing on conjunction with an Oral Irrigator or toothbrushing without an Oral Irrigator (N=15/treatment). Subjects will be instructed to brush twice a day for approximately three (3) weeks with their assigned products and return for plaque and gingivitis measures at approximately three (3) weeks after the Baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and receive a copy of the signed Informed Consent form;
* Be at least 18 years of age;
* Typically use a manual toothbrush;
* Be in good general health as determined by the investigator/designee based on a review/update of their medical history;
* Possess a minimum of 16 scorable teeth (excluding third molars) with facial and lingual scorable surfaces;
* Have a Baseline MGI score between 1.75 and 2.5;
* Have a Baseline TQHPI score of at least 2.00;
* Have a Baseline between 20 and 80 Bleeding sites;
* Abstained from all oral hygiene procedures for approximately 12 hours prior to this visit and agree to do the same prior to the subsequent visit;
* Abstained from eating, drinking*, chewing gum and using tobacco for at least 4 hours prior to this visit and agree to do the same prior to the subsequent visit. *(Exception: Allowed small sips of water up until 45 minutes prior to their appointment time.)
* Agree not to participate in any other oral care study for the duration of this study;
* Agree to delay any elective dentistry, including dental prophylaxis, and to report any non-study dentistry received during the course of this study;
* Agree to refrain from using any non-study toothbrushes, dentifrices, mouth rinses, tooth whitening products or floss for the study duration; and
* Agree to return for their scheduled visits and to follow all study procedures.

Exclusion Criteria:

* Hypersensitivity to dyes;
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* Any carious lesions requiring restorative treatment;
* Active treatment for periodontitis;
* Any fixed facial orthodontic appliances or retainers;
* Use of any antibiotic medication or a prescription mouth rinse any time within the 2 weeks prior to study initiation; or
* Any disease or conditions that could be expected to interfere with examination; procedures or the subject safely completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Regimen | Control Regimen
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Regimen | Control Regimen | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (15.61) | 49.2 (13.04) | 48.2 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: MGI-Modified Gingival Index
Description: Modified Gingival Index score after 3 weeks of product use. Gingivitis will be scored on the buccal and lingual marginal gingival and interdental papilla of all scorable teeth (six scores per tooth):0 = normal (absence of inflammation); 1 = mild inflammation (slight change of color, little change in texture) of any portion of the gingival unit; 2 = mild inflammation of the entire gingival unit; 3 = moderate inflammation (moderate glazing, redness, edema and/or hypertrophy) of the gingival unit; 4 = severe inflammation (marked redness and edema/hypertrophy, spontaneous bleeding or ulceration) of the gingival unit. MGI whole mouth score is computed by summing the scores and dividing by the number of scorable sites examined.
Time Frame: MGI Score after 3 weeks of product use.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Regimen | Control Regimen
Number analyzed (Participants) | 15 | 15
score on a scale | 0.30 (0.081) | -0.13 (0.047)

2. Primary Outcome: GBI-Gingival Bleeding Index
Description: Gingival Bleeding Index score after 3 weeks of product use. Each of the 3 gingival areas, i.e., buccal, mesial/dystal and lingual, of the teeth will be probed in this manner waiting approximately 30 seconds before recording the number of gingival units which bleed, according to the following scale: 0 = absence of bleeding after 30 seconds; 1 = bleeding observed after 30 seconds; 2 = immediate bleeding observed. GBI whole mouth score is computed by summing the scores and dividing by the number of scorable sites examined.
Time Frame: GBI score after 3 weeks of product use.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Regimen | Control Regimen
Number analyzed (Participants) | 15 | 15
score on a scale | 0.16 (0.017) | -0.06 (0.030)

3. Secondary Outcome: Plaque- TMQHP
Description: Turesky Modified Quigley-Hein Plaque Index score after 3 weeks of product use. The plaque deposits on the buccal, lingual, and whole mouth average plaque scores will be calculated for each subject and tooth surfaces by totaling the scores and dividing by the number of gradable sites examined. Scoring criteria are shown below. 0=No Plaque; 1=Separate flecks of plaque at the cervical margin; 2=A thin, continuous band of plaque (up to 1 mm) at the cervical margin; 3=A band of plaque wider than 1mm, but covering less than one third of the side of the crown of the tooth; 4=Plaque covering at least one third, but less than two thirds of the side of the crown of the tooth; 5=Plaque covering two thirds or more of the side of the crown of the tooth; 8=Ungradable site; 9=Missing tooth
Time Frame: TMQHP score after 3 weeks of product use.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Regimen | Control Regimen
Number analyzed (Participants) | 15 | 15
score on a scale | 0.28 (0.038) | 0.10 (0.048)

ADVERSE EVENTS:
Time Frame: after 3 weeks of product use
Arm/Group | Test Regimen | Control Regimen
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT04899440/Prot_SAP_000.pdf